CLINICAL TRIAL: NCT03781791
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate Safety, Tolerability and Efficacy of Orally Administered ENT-01 for the Treatment of Parkinson's Disease-Related Constipation (KARMET)
Brief Title: Orally Administered ENT-01 for Parkinson's Disease-Related Constipation (KARMET)
Acronym: KARMET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Enterin Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ENT-01-030
Record Dates: First submitted 2018-11-27; First posted 2018-12-20 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-01

CONDITIONS: Constipation; Parkinson Disease
MeSH Terms: conditions — Constipation; Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental): ENT-01 tablet will be taken once daily by mouth.
  Interventions: Drug: Active Investigational Treatment ENT-01
- Placebo Treatment (Placebo Comparator): Placebo tablet will be taken once daily by mouth.
  Interventions: Drug: Placebo Treatment

INTERVENTIONS:
Drug: Active Investigational Treatment ENT-01 — ENT-01 will be administered in tablet form, once daily.
  Other Names: ENT-01
  Arms: Active Treatment
Drug: Placebo Treatment — Placebo will be administered in tablet form, once daily.
  Arms: Placebo Treatment

SUMMARY:
This study will be conducted as a multi-center, randomized, double-blind, placebo-controlled study. Approximately 72 patients will be randomized 3:1 to treatment or placebo, with approximately 54 patients allocated to receive the active investigational product and approximately 18 patients allocated to receive placebo.

- Study Update-

Amendment 3 - In this amendment, an additional 80 patients (approximately) will be randomized 1:1 to treatment or placebo (double-blind) with approximately 40 subjects allocated to each group.

DETAILED DESCRIPTION:
The study will be conducted on an out-patient basis. Each patient will have 6 visits to the clinic: a screening visit, a randomization visit, 3 follow up visits, and 1 end of study visit.

Patient randomization will be stratified based upon the baseline weekly complete spontaneous bowel movement rate (CSBM) established during the screening period. Patients will be allowed to adjust their dosing, based upon protocol specifications. Rescue medications will be provided to all patients to ensure they move their bowels on a regular basis.

Patients will also be asked to participate in up to 2 sub-studies: a pk study and/or a stool microbiome study. The first 20 patients to consent to the pk study will have additional blood samples taken at randomization and at 2 follow up visits. The first 20 patients to consent to the stool microbiome study will provide stool samples at randomization and at 2 follow up visits.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects aged 30-90 years, both genders
2. Subjects must provide written informed consent and be willing and able to comply with study procedures.
3. Subjects must be diagnosed with Parkinson's Disease defined as the presence of at least three of the following cardinal features, in the absence of alternative explanations or atypical features: rest tremor, rigidity, bradykinesia and/or akinesia, postural and gait abnormalities.
4. There are insufficient criteria for Irritable Bowel Syndrome (IBS)
5. Constipation which has been present for over 6 months and is unresponsive to first line, typically over the counter treatments such as Milk of Magnesia (1g), Miralax (17g in 8 ounces of water) or the equivalent at least once weekly with an inconsistent response over a 6-week period or the subject is dissatisfied with first line treatments.
6. Body mass index (BMI) of 18-40 kg/m2
7. Subjects must fulfill Rome IV criteria for functional constipation which includes 2 or more of the following:

   1. Straining during at least 25% of defecations
   2. Lumpy or hard stools in at least 25% of defecations
   3. Sensation of incomplete evacuation for at least 25% of defecations
   4. Sensation of anorectal obstruction/blockage for at least 25% of defecations
   5. Manual maneuvers to facilitate at least 25% of defecations (e.g., digital evacuation, support of the pelvic floor)
8. Self-report of fewer than 3 complete spontaneous bowel movements per week
9. Loose stools are rarely present without the use of laxatives
10. Subjects must be able to read, understand, and accurately record data into the diary to guarantee full participation in the study.
11. Female subjects must have negative serum or urine pregnancy tests and must not be lactating. For females able to bear children, a hormonal (i.e., oral, implantable, or injectable) and single-barrier method, or a double-barrier method of birth control must be used throughout the study. A vasectomized partner will be allowed as one in conjunction with another single-barrier method.
12. Female subjects unable to bear children must have this documented in the CRF (i.e., tubal ligation, hysterectomy, or postmenopausal [defined as a minimum of one year since the last menstrual period]). Post-menopausal status will be confirmed by follicle stimulating hormone (FSH) in women less than 60 years of age.

Exclusion Criteria:

1. Unable or unwilling to provide informed consent or to comply with study procedures.
2. Diagnosis of secondary constipation beyond that of Parkinson's Disease
3. Review of Screening Diaries indicates fewer than 11 days of diary completion and/or 3 or more complete spontaneous bowel movements (CSBM) per week based upon the average CSBM rate reported during the Screening Period
4. A compromised gastrointestinal system which includes:

   1. Structural, metabolic, or functional GI diseases or disorders
   2. Acute GI illness within 2 weeks of the screening visit
   3. History of major GI surgery within 30 days of the screening visit (a history of cholecystectomy, polypectomy, hernia repair or appendicectomy are not exclusionary as long as they were performed more than 30 days before the screening visit)
5. Unable or unwilling to withdraw from laxatives, opiates, clonazepam, or any medications which may cause constipation, 2 weeks prior to the dose adjustment period and throughout the rest of the study.
6. Unable or unwilling to withdraw from proton pump inhibitors and antacids at the end of the screening period.
7. Unable or unwilling to withdraw from pimavanserin during the study.
8. Any clinically significant abnormalities on screening laboratories or physical examination requiring further evaluation or treatment.
9. Neurological disorder other than Parkinson's Disease that in the opinion of the investigator might interfere with the conduct of the study.
10. On treatment with intra-jejunal dopamine or carbidopa/levodopa (i.e. Duopa).
11. Subjects starting a new Parkinson's Disease medication or modifying an existing medication within 2 weeks prior to enrollment.
12. Unable to maintain a stable diet regimen.
13. Subjects with a cognitive impairment that preclude them from understanding the informed consent.
14. Subjects placed under legal guardianship.
15. Females who are pregnant or breastfeeding.
16. History of excessive alcohol use or substance abuse.
17. Participation in an investigational drug trial within the month prior to dosing in the present study.
18. Any other reason, which, in the opinion of the investigator, would confound proper interpretation of the study.

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2021-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zasloff, MD PhD, Study Chair — Enterin Inc.; Denise Barbut, MD, FRCP, Study Director — Enterin Inc.
Locations (51):
- United States (51):
  - Banner Sun Health Research Institute, Sun City, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Neuro Pain Medical Center, Fresno, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - SC3 Research - Pasadena, Pasadena, California
  - Trial Connections - Care Access Research, Santa Clarita, Santa Clarita, California
  - Rocky Mountain Movement Disorders Center, Englewood, Colorado
  - Associated Neurologist of Southern CT, Fairfield, Connecticut
  - Care Access Research, Norwich, Norwich, Connecticut
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - JEM Research Institute, Atlantis, Florida
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - Elias Research - Floridian Research Institute, Miami, Florida
  - Elias Research - Allied Biomedical Research Institute, Miami, Florida
  - Pharmax Research of South Florida, Miami, Florida
  - MEDSOL Clinical Research, Port Charlotte, Florida
  - Parkinson's Disease Treatment Center of SWFL, Port Charlotte, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Palm Beach Neurology and Premier Research Institute, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - BTC Network - Community Clinical Research Center, Anderson, Indiana
  - Interspond - The Neuromedical Clinic of Central Louisiana, Alexandria, Louisiana
  - The NeuroMedical Center, P.C., Baton Rouge, Louisiana
  - Parkinson's and Movement Disorders Center of Maryland, Elkridge, Maryland
  - Henry Ford West Bloomfield Hospital, West Bloomfield, Michigan
  - Neurology Associates Clinical Research, Lincoln, Nebraska
  - Interspond - Neurology Center of Las Vegas, Las Vegas, Nevada
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Evolution Research Group - Neuroscience Research Institution, Toms River, New Jersey
  - Neuroscience Researc Institute of NJ, Toms River, New Jersey
  - Albany Medical College, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest Baptist Medical Center, Wake Forest, North Carolina
  - Dayton Center for Neurological Disorders, Centerville, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Elias Research - Neurology Diagnostics Research, Dayton, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Penn State University, Hershey, Pennsylvania
  - Interspond - Premier Neurology, Greer, South Carolina
  - Interspond - Metrolina Neurological Associates, Old Point Station, South Carolina
  - North Texas Movement Disorders Institute, Bedford, Texas
  - BTC Network - Neurological Associates of North Texas, Dallas, Texas
  - Clinical Trial Network, Houston, Texas
  - Sentara Neuroscience Institute, Norfolk, Virginia
  - Evergreen Health - Booth Gardner Parkinson's Care Center, Kirkland, Washington
  - University Physicians & Surgeons, Inc. dba Marshall Health, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Camilleri M, Subramanian T, Pagan F, Isaacson S, Gil R, Hauser RA, Feldman M, Goldstein M, Kumar R, Truong D, Chhabria N, Walter BL, Eskenazi J, Riesenberg R, Burdick D, Tse W, Molho E, Robottom B, Bhatia P, Kadimi S, Klos K, Shprecher D, Marquez-Mendoza O, Hidalgo G, Grill S, Li G, Mandell H, Hughes M, Stephenson S, Vandersluis J, Pfeffer M, Duker A, Shivkumar V, Kinney W, MacDougall J, Zasloff M, Barbut D. Oral ENT-01 Targets Enteric Neurons to Treat Constipation in Parkinson Disease : A Randomized Controlled Trial. Ann Intern Med. 2022 Dec;175(12):1666-1674. doi: 10.7326/M22-1438. Epub 2022 Nov 8. PMID 36343348

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Active Treatment | Placebo Treatment
Started | 93 | 57
Completed | 67 | 50
Not Completed | 26 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Treatment | Placebo Treatment | Total
Number analyzed (Participants) | 93 | 57 | 150
Age, Continuous [Median (Standard Deviation); unit: years] | 67.0 (8.75) | 71.0 (6.66) | 69.0 (8.09)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 25 | 63
  Male | 55 | 32 | 87
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 87 | 52 | 139
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 93 | 58 | 151
Years of Constipation [Mean (Standard Deviation); unit: years] | 10.2 (10.94) | 16.4 (19.73) | 12.6 (15.2)

OUTCOME MEASURES:

1. Primary Outcome: The Number of Participants Who Experience Treatment Related Adverse Events-Safety Endpoint
Description: The number of treatment related adverse events as reported and assessed by NCI CTCAE v.4.3.
Time Frame: Through Study treatment up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 93 | 57
Participants | 44 | 7

2. Primary Outcome: The Number of Participants Who Experience Dose Limiting Toxicity Adverse Events
Description: The number of participants who experience dose limiting toxicity adverse events as reported and assessed by NCI CTCAE v.4.3.
  Per protocol, dose limiting toxicity adverse events are vomiting, diarrhea, abdominal pain and dizziness.
Time Frame: Through Study treatment Dosing Period up to 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 93 | 57
Participants | 38 | 4

3. Primary Outcome: Change in Baseline Weekly CSBM-Primary Efficacy Endpoint
Description: Change from participant's weekly CSBM baseline rate during treatment fixed Dose period.
  The fixed dose period begins on the first day or the subject's highest dose at which the subject did not experience a dose limiting toxicity (nausea, vomiting, diarrhea or dizziness) The fixed dose period will not be a specific time period for all subjects since each subject will start the fixed dose period based on their tolerability to ENT-01 dosing.
Time Frame: 25 day treatment period, part of which is at a fixed dose.
Measure: Mean (Standard Deviation); unit: spontaneous movements per week
Arm/Group | Active Treatment | Placebo Treatment
Number analyzed (Participants) | 93 | 57
spontaneous movements per week
  Baseline | 1.1 (1.01) | 1.0 (1.05)
  Fixed Dose Period | 3.9 (3.43) | 2.3 (2.49)

ADVERSE EVENTS:
Time Frame: Adverse events are collected once ICF signed through 30 post last dose of study medication (approximately 10 weeks plus 30 days post dose follow-up)
Arm/Group | Active Treatment | Placebo Treatment
All-Cause Mortality (participants affected / at risk) | 0/93 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/93 | 0/57
Other Adverse Events (participants affected / at risk) | 61/93 | 10/57
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Active Treatment (N=93) | Placebo Treatment (N=57)
Vomiting (Gastrointestinal disorders) | 7 | 0
Diarrhoea (Gastrointestinal disorders) | 18 | 3
Abdominal Pail (Gastrointestinal disorders) | 7 | 3
Nausea (Gastrointestinal disorders) | 32 | 3
Dizziness (Nervous system disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-17): https://cdn.clinicaltrials.gov/large-docs/91/NCT03781791/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT03781791/SAP_001.pdf